CLINICAL TRIAL: NCT04941144
Title: General Use Results Survey: Spikevax Intramuscular Injection (Previously COVID-19 Vaccine Moderna Intramuscular Injection) During the Early Phase of Treatment With Novel Corona Vaccine, Follow-up of Key Survey Participants
Brief Title: Long-Term Follow-up Survey of COVID-19 Vaccine After Vaccination
Status: Completed | Type: Observational
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: mRNA-1273-P918; jRCT2031210168 (Registry Identifier: jRCT)
Record Dates: First submitted 2021-06-25; First posted 2021-06-28 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Coronavirus Disease (COVID-19)
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- COVID-19 Vaccine Intramuscular Injection 0.5 milliliters (mL): COVID-19 vaccine intramuscular injection, 2 doses of 0.5 mL per dose administered intramuscularly at an interval of 4 weeks.
  Interventions: Biological: COVID-19 Vaccine

INTERVENTIONS:
Biological: COVID-19 Vaccine — COVID-19 Vaccine Intramuscular Injection
  Other Names: COVID-19 Vaccine Moderna Intramuscular Injection; Spikevax Intramuscular Injection

SUMMARY:
This study is a long-term follow-up survey of Japanese people after their second vaccination with the Moderna COVID-19 vaccine.

The study sponsor will not be involved in how the participants are treated but will provide instructions on how the clinics will record what happens during the study.

The main aim of the study is to check for long-term side effects of the COVID-19 vaccine. This will be from 28 days to 12 months after the second vaccination of the COVID-19 vaccine.

The number of visits to the clinic will depend on the clinic's standard practice.

ELIGIBILITY:
Inclusion Criteria:

Participants who have participated in the preceding cohort study and has subsequently provided written consent to participate in this study.

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The population of this survey are vaccinated participants who meet the inclusion/exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 8538 (Actual)
Dates: Start 2021-12-22 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Serious Adverse Events (SAE) | 11 months (From 28 days to 12 months after the second vaccination)
  An SAE is defined as any untoward medical occurrence that: Results in death, Is life-threatening, Requires in patient hospitalization or prolongation of existing hospitalization, Results in persistent or significant disability/incapacity, Leads to a congenital anomaly/birth defect in the offspring of a participant, or Is an important medical event.

SECONDARY OUTCOMES:
Number of Participants who Take COVID-19 Pathogen (Severe Acute Respiratory Syndrome coronavirus [SARS-CoV-2]) Test during the Study | 11 months (From 28 days to 12 months after the second vaccination)
Number of Participants who Developed COVID-19 during the Study | 11 months (From 28 days to 12 months after the second vaccination)
Number of Participants Who Have Severe COVID-19 Infection during the Study Evaluated by Investigator | 11 months (From 28 days to 12 months after the second vaccination)
  Number of participants who have severe COVID-19 infection during the study evaluated by investigator will be reported. Investigator will evaluate the severity of COVID-19 infection with COVID-19 information entered in the case report form in reference to "Guidance for Clinical Practice of Novel Coronavirus Infection (COVID-19)".

CONTACTS AND LOCATIONS:
Locations (1):
- Moderna selected site, Tokyo, Japan